CLINICAL TRIAL: NCT06177613
Title: Advantages of Early Intrauterine Transfer of "Blank" Culture Medium Prior to 1st or 2nd Transfer of Thawed Embryo(s). Randomized, Single-blind, Multicenter Controlled Trial.
Brief Title: Advantages of Early Intrauterine Transfer of "Blank" Culture Medium Prior to 1st or 2nd Transfer of Thawed Embryo(s).
Acronym: TRABLAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PHRC-I/2022/NR-01
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Single Embryo Transfer; Fertilization in Vitro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With blank culture (Experimental)
  Interventions: Procedure: Blank culture transfer
- Without blank culture (Sham Comparator)
  Interventions: Procedure: Sham transfer

INTERVENTIONS:
Procedure: Blank culture transfer — A maximum of 0.1 ml of gassed embryo culture medium preheated to 37°C is injected into the uterine cavity transcervically using an embryo transfer catheter placed just beyond the internal os, two to 3 days before transfer of the thawed embryo
  Arms: With blank culture
Procedure: Sham transfer — An intermediate transfer step is added two or three days before the planned transfer of the frozen embryo but with an empty catheter.
  Arms: Without blank culture

SUMMARY:
Despite technical advances in Medically Assisted Reproduction (AMP), the success of fertility treatments is sometimes limited by embryo implantation failure. The coordinated development of the embryo and the uterine endometrium requires close communication between the maternal tissue and the embryo. In in vitro fertilization (IVF), embryo transfer generally takes place between the 2nd (D2) and the 6th (D6) day following oocyte fertilization. Recent studies have shown the advantages of sequential transfer (transfer of an embryo on D2/D3 followed by the transfer of another embryo on D5/D6), with higher implantation and clinical pregnancy rate, fewer miscarriages, more live births, and yet no increase in multiple pregnancies. However, the American Society for Reproductive Medicine recommendations continue to prioritize the transfer of a single embryo for all patients aged under 38. To improve pregnancy rates for patients having a single embryo transferred, the study investigators wish to carry out on "blank" transfer, based on the principle of sequential transfer. The study investigators hypothesize that a culture medium, placed in the uterus before the time of embryo transfer, will modify immune tolerance. The study will test whether transferring the same culture medium in an equivalent quantity as during the real transfer into the uterus 2/3 days before the embryo transfer will improve tolerance to this foreign medium and, therefore, embryo implantation. The aim of this study is thus to evaluate the impact of a "blank" transfer with culture medium alone, on the results of frozen embryo transfers (FET) from IVF.

ELIGIBILITY:
Inclusion Criteria:

* Having had a first "fresh" or frozen embryo transfer, whatever the embryo's stage of development, transfer followed by pregnancy failure ;
* Frozen embryos must be at least D3 stage;
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice or state guardianship

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1154 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinically progressive pregnancy rate between groups | 12 weeks of amenorrhea
  Measured on first-trimester ultrasound

SECONDARY OUTCOMES:
Occurrence of pregnancy between groups | Day 14
  Defined by a positive beta HCG test ≥ 100 IU/ml
Occurrence of a biochemical pregnancy between groups | Day 14
  Defined by a positive beta HCG test ≥ 10 IU/ml and < 100 IU/ml
Occurrence of a clinical pregnancy between groups | 6 weeks of amenorrhea
  Defined by a positive beta HCG test ≥ 100 IU/ml and presence of at least one gestational sac on dating ultrasound
Occurrence of an early miscarriage between groups | 12 weeks of amenorrhea
  Defined by the presence of a pregnancy defined by a positive beta HCG test ≥ 100 IU at D14 and the absence of an evolving clinical pregnancy at first-trimester ultrasound
Occurrence of live birth | Upon giving birth (maximum month 9)
  Yes/no
Differential cost-result ratio | End of study (Year 3)
  Ratio of the cost differential and the number of additional live births (additional progressive clinical pregnancies) between the two strategies, to evaluate the cost per additional live birth.
Total estimated expenditure for the two care strategies compared (budget impact analysis) over a one-year time horizon. | End of study (Year 3)
  Calculated at national level (implementation of the system and consumption of care)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Rougier, Principal Investigator — CHU de Nimes
Locations (7):
- France (6):
  - Hôpital Antoine Béclère, Clamart
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - CHU Arnaud de Villeneuve, Montpellier
  - Clinique Saint Roch, Montpellier
  - CHU de Nîmes, Nîmes
  - Clinique Saint-Pierre, Perpignan
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No